CLINICAL TRIAL: NCT03995875
Title: Real World Evidence of Long-term Safety and Efficacy in Patients Treated With Durvalumab After Concurrent Chemoradiation for Unresectable Stage III NSCLC.
Acronym: AYAME
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Japan Lung Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: D4194R00013
Record Dates: First submitted 2019-06-06; First posted 2019-06-24 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC, stageIII, Durvalumab, Japanese, Real world
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No

SUMMARY:
This observational study is designed to assess the long term safety of the durvalumab treatment period including subsequent treatment period and demonstrate the efficacy of patients treated with durvalumab following chemoradiation therapy in the real world.

DETAILED DESCRIPTION:
Study design: Prospective multi-center non-interventional cohort study Data Source(s): Medical records of patients who are treated with durvalumab following chemoradiation therapy Study Population: Patients prescribed and treated with durvalumab for unresectable stage III non-small cell lung cancer (NSCLC) at first time following chemoradiation therapy and who provide written informed consent.

Exposure(s): durvalumab Outcome(s): Summary of pneumonitis and adverse event special interest (AESI), progression free survaival (PFS), overall survaival (OS), Reasons of discontinuation of durvalumab treatment, Details of subsequent treatments after durvalumab Sample Size Estimations: 500 patients Statistical Analysis: Only descriptive analysis and no formal test

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive durvalumab for unresectable stage III NSCLC at first time following chemoradiation therapy.
* Patients who provided written informed consent.

Exclusion Criteria:

* Patients who would join Post Marketing Surveyllance for durvalumab.
* Patients who would join any interventional clinical studies using unapproved drugs or off-label use of drugs from first diagnosis to the end of the durvalumab treatment
* Age < 20

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Total 500 patients who receive durvalumab for unresectable stage III NSCLC at first time following chemoradiation therapy will be enrolled. The patients should be registered consecutively in each site.
Sampling Method: Non-Probability Sample
Enrollment: 529 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Incidence of pneumonitis and AESI | 3 years
  Pneumonitis and AESIs will be summarized at least following categories
  * Pneumonitis within three years from the start of durvalmab treatment
  * Pneumonitis and AESIs during treatment period of durvalmab
  * Pneumonitis and AESIs after durvalmab treatment
To assess progression free survival (PFS) of durvalumab | PFS is assessed as PFS median for time of 3 years
  PFS is defined as the time from the start of durvalumab treatment to first progression disease (PD) or death, whichever is earlier. In case the patients without progression or death, patients will be censored at the last follow-up date or the first date of the 1st subsequent treatment, whichever is earlier.

SECONDARY OUTCOMES:
To assess overall survaival (OS) of durvalumab | OS is assessed as median OS for time of 3 years
  OS is defined as the time from the date of start of the durvalumab treatment until death due to any causes. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
Incidence of pneumonitis and AESIs in patient subset populations | 3 years
  Summary of pneumonitis and AESIs in each durvalumab treatment status in patient subset populations

CONTACTS AND LOCATIONS:
Locations (43):
- Japan (43):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Toyoake, Aichi-ken
  - Research Site, Matsuyama, Ehime
  - Research Site, Kurume, Fukuoka
  - Research Site, Maebashi, Gunma
  - Research Site, Asahikawa, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Akashi, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Kasama, Ibaraki
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Morioka, Iwate
  - Research Site, Sagamihara, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Matsubara, Mie-ken
  - Research Site, Natori-shi, Miyagi
  - Research Site, Sendai, Miyagi
  - Research Site, Nishihara, Okinawa
  - Research Site, Hirakata, Osaka
  - Research Site, Sakai, Osaka
  - Research Site, Sayama, Osaka
  - Research Site, Hidaka, Saitama
  - Research Site, Izumo, Shimane
  - Research Site, Mishima, Shizuoka
  - Research Site, Mibu, Tochigi
  - Research Site, Shimotsuke, Tochigi
  - Research Site, Bunkyo, Tokyo
  - Research Site, Chūō, Tokyo
  - Research Site, Koto, Tokyo
  - Research Site, Mitaka, Tokyo
  - Research Site, Shinjuku, Tokyo
  - Research Site, Iwakuni, Yamaguchi
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Kyoto
  - Research Site, Nagasaki
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Saitama
  - Research Site, Tokushima
  - Research Site, Wakayama

REFERENCES:
- [Derived] Kenmotsu H, Saito Y, Ninomiya K, Uematsu S, Akdemir B, Fukui A, Koto R, Fujiwara M, Iwao C, Kitagawa H, Yoshino I, Gemma A, Mitsudomi T, Yamamoto N. Long-Term Safety and Effectiveness of Durvalumab in Unresectable Stage III NSCLC in Japan: A Multicenter Prospective Study (AYAME). J Thorac Oncol. 2025 Aug 18:S1556-0864(25)01014-7. doi: 10.1016/j.jtho.2025.08.010. Online ahead of print. PMID 40835220
- See also: CSR Synopsis AYAME study — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4194R00013&attachmentIdentifier=4733ff81-2c99-433b-96f7-03136b7d8f3b&fileName=AYAME_study_CSR_synopsis_version1.0_20241119_redacted.pdf&versionIdentifier=